CLINICAL TRIAL: NCT07397455
Title: Development of a Controlled Human Infection Model for Assessment of SARS-CoV-2 Omicron Subvariants
Acronym: COVHIC003
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 172082
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: SARS-CoV-2 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Dose Escalation/Expansion design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1a: SARS-CoV-2 Omicron EG.5.1 (Experimental): Starting dose 10^5 TCID50, vaccinated, pre-selection for low serum antibodies, n = up to 12
  Interventions: Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^5 TCID50
- Group 1b: SARS-CoV-2 Omicron EG.5.1 (Experimental): Dose escalate: 10^6 TCID50, vaccinated, pre-selection for low serum antibodies, n = up to 12
  Interventions: Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^6 TCID50
- Group 1c: SARS-CoV-2 Omicron EG.5.1 (Experimental): Dose de-escalate: 10^4 TCID50, vaccinated, pre-selection for low serum antibodies, n = up to 12
  Interventions: Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^4 TCID50
- Group 2: SARS-CoV-2 Omicron EG.5.1 (Experimental): 10^6 TCID50 with multiple doses and/or lower sero-screening threshold
  Interventions: Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^6 TCID50

INTERVENTIONS:
Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^5 TCID50 — 10^5 TCID50
  This is a SARS-CoV-2 Omicron EG.5.1 challenge agent which has not been given in controlled human infection studies previously.
  Arms: Group 1a: SARS-CoV-2 Omicron EG.5.1
Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^6 TCID50 — 10^6 TCID50 This is a SARS-CoV-2 Omicron EG.5.1 challenge agent which has not been given in controlled human infection studies previously
  Arms: Group 1b: SARS-CoV-2 Omicron EG.5.1; Group 2: SARS-CoV-2 Omicron EG.5.1
Biological: SARS-CoV-2 Omicron EG.5.1 challenge agent 10^4 TCID50 — 10^4 TCID50
  This is a SARS-CoV-2 Omicron EG.5.1 challenge agent which has not been given in controlled human infection studies previously
  Arms: Group 1c: SARS-CoV-2 Omicron EG.5.1

SUMMARY:
COVHIC003 is a human infection challenge study in which healthy adults aged 18-50 previously vaccinated with an approved COVID-19 vaccine will be administered a SARS-CoV-2 Omicron EG.5.1 variant given by drops in the nose. The aim is to achieve breakthrough upper-respiratory infection in a proportion of volunteers with mild or no illness, providing information on the course of Omicron infection and the immune response in vaccinated people. This study will establish an optimised challenge dose and model that can then be used to evaluate new vaccines and treatments in follow-on trials. Participants will stay in a quarantine unit for approximately 10-12 days, depending on infection status, and will be closely monitored with regular swabs, blood tests and symptom assessments throughout their stay. They will be followed up by the study team for 6 months after being discharged. This study is sponsored by Imperial College London and forms part of the MUSICC project which is led by Imperial College London and co-funded by the European Union's Horizon Europe Programme and the Coalition for Epidemic Preparedness Innovations (CEPI). Quarantine will take place at specialist facilities in Oxford or at the Royal Free Hospital in London.

ELIGIBILITY:
Inclusion Criteria:

* The study informed consent form has been signed and dated by the participant and the Investigator
* Adults age between 18 and 50 years inclusive (at the time of enrolment)
* Evidence of having had at least one COVID-19 vaccine, with the last vaccination at least 3 months before enrolment
* Positive serology for SARS-CoV-2 at (pre)screening
* Sero-suitable as defined by having serum and/or nasal antibody titres less than a pre-defined cut-off of a defined assay(s) which will be specified in a separate SOP and based on accumulating antibody data
* People of child-bearing potential (POCBP) must be willing and able to use contraception as described in the study protocol from 2 weeks before the scheduled date of viral challenge until the end discharge from quarantine.

Negative urine pregnancy tests will be required at screening and on day 0 prior to inoculation. On admission to the quarantine unit a negative serum beta human chorionic gonadotropin (β-hCG) is required

* Male participants who are willing to use one of the contraception methods described in the study protocol, from the time of the date of viral challenge until the end of quarantine
* Agree to abstain from sexual activity or use effective contraception from the start of treatment with Paxlovid until 7 days after completing treatment with Paxlovid should they receive it
* In good health with no history of clinically significant medical conditions (as described in Exclusion criteria) that would interfere with participant safety, as defined by medical history, physical examination and routine laboratory tests, ECG, and Chest X-Ray and determined by the Investigator at an admission evaluation
* Participants will have a documented medical history either prior to entering the study and/or following medical history review with the study physician at screening
* Willing to be registered with The Over-Volunteering Protection Service (TOPS)
* Willing and able to commit to participation in the study.

Exclusion Criteria:

* History or evidence of any clinically significant or currently active cardiovascular, (including thromboembolic events), respiratory, dermatological, gastrointestinal, endocrine, haematological, hepatic, immunological, rheumatological, metabolic, urological, renal, neurological, psychiatric illness
* Any significant abnormality altering the anatomy or function of the nose or nasopharynx in a substantial way (including loss of or alterations in smell or taste), a clinically significant history of epistaxis (large nosebleeds) within the last 3 months, nasal or sinus surgery within 6 months of inoculation
* Clinically-active, symptomatic rhinitis (including hay fever) or history of severe rhinitis, or seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine
* History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food or drug, as assessed by the Investigator
* Significant history or presence of drug or alcohol misuse (exceeding >28 units a week)
* Current use of any drugs taken through the nasal or inhaled route including recreational drugs
* Psychiatric illness including participants with a history of depression and/or anxiety with associated severe psychiatric comorbidities, for example psychosis.
* Current active smokers, equivalent to >5 cigarettes per week, including use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch) or electronic cigarettes. • Participants who have smoked ≥5 pack years at any time [5 pack years is equivalent to one pack of 20 cigarettes a day for 5 years]) or the equivalent amount of nicotine if using alternative forms. • Ex-smokers who have smoked <5 pack years at any time must not of have regularly smoked in the last 3 months equivalent to >5 cigarettes per week.
* Family history of 1st degree relative aged 50 years or less with sudden cardiac or unexplained death
* Personal or Family History of unexpectedly severe COVID-19, adverse response to any other viral disease e.g. Guillain-Barré, or a family history (described as a 1st degree relative) with clotting disorders
* A total body weight of ≤ 45kg and a Body Mass Index (BMI) ≤18 kg/m2 and ≥28 kg/m2. The upper limit of BMI may be increased to ≤ 30kg/m2 at the Investigator's discretion, in the case of physically fit muscular individual
* Venous access deemed inadequate for the phlebotomy demands of the study.
* Any clinically significant abnormal finding on screening biochemistry, haematology and microbiology blood tests or urinalysis i.e. grade 1 lab abnormalities or above apart from minor deviations which are clinically acceptable and approved by the Investigator
* A forced expiratory volume in 1 second (FEV1) and a forced vital capacity (FVC) <80% of predicted value calculated using ATS/ERS guidance. Spirometry will be performed only if the mMRC dyspnoea score ≥1 or if clinically indicated
* Twelve-lead ECG recording with clinically relevant abnormalities as judged by the Investigator
* History of, or currently active symptoms suggestive of upper or lower respiratory tract infection (including reduced sense of taste and smell, raised body temperature and/or persistent cough) within 4 weeks prior to viral challenge
* Presence of cold-like symptoms and/or fever (defined as participant presenting with a temperature reading of >37.9ºC) on Day -2, Day -1 and/or pre-challenge on Day 0.
* Evidence of any respiratory pathogens (on Respiratory PCR from upper respiratory tract sample) prior to challenge virus inoculation on admission to the quarantine unit
* Evidence of a live vaccine within 60 days prior to the planned date of viral challenge, a non-live vaccine within 30 days prior to the planned date of viral challenge or intention to receive any vaccination(s) before the day 28 follow-up visit. (NB. No travel restrictions applied after the Day 28 Follow-up visit).
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned date of viral challenge or planned during the 3 months after the final visit.
* Medications

  1. Use of any medication or product (prescription or over-the-counter), for symptoms of hay fever, nasal congestion or respiratory tract infections or dermatitis/eczema including the use of regular nasal or medium-high potency dermal corticosteroids, antibiotics and First Defence™ (or generic equivalents) within 7 days prior to the planned date of viral challenge apart from those described in Table 7, Permitted Medication or agreed by the Investigator.
  2. Receipt of any investigational drug within 3 months prior to the planned date of viral challenge.
  3. Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge.
  4. Receipt of systemic (intravenous and/or oral) glucocorticoids or antiviral drugs known to have activity against respiratory viruses within 6 months prior to the planned date of viral challenge (excluding Pre-Exposure Prophylaxis (PrEP)).
  5. Over the counter medications (e.g., paracetamol or ibuprofen) where the dose taken over the preceding 7 days prior to the planned date of viral challenge had exceeded the maximum permissible 24-hour dose (e.g., >4g per day of paracetamol over the preceding week).
  6. Chronically used medications, including any medication known to be a moderate/potent inducer or inhibitor of cytochrome P450 enzymes, within 21 days prior to the planned date of viral challenge, except for those agreed by the Investigator.
  7. Participants who have received any systemic chemotherapy agent, immunoglobulins, or other cytotoxic or immunosuppressive drugs at any time.
  8. Concurrent use of medications strongly contraindicated for use with Paxlovid unless confirmed alternative rescue therapy will be available to the site at the time of enrolment
* Prior participation in another human viral challenge study in the preceding 6 months taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study. The participant must also have completed the follow up visit requirements of the previous viral challenge study
* Any invasive nasal sampling procedure in the month before date of expected viral challenge in this study (excluding study tolerance test or routine tests for COVID-19)
* Participant is mentally or legally incapacitated in the opinion of the Investigator
* POCBP who:

  1. Are breastfeeding within 6 months of study commencement, or
  2. Had been pregnant within 6 months prior to the study, or
  3. Had a positive pregnancy test at any point during screening or prior to inoculation with challenge virus
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 2 years, the elderly (>65 years), immunosuppressed persons, or those with chronic respiratory disease
* Anyone who works on the study (e.g. a delegated study nurse) or in close proximity to the study at the sponsor organisation, participating trial sites or any contract research organisations involved in this study.
* Anyone who is first degree related to, or resides with, anyone who is a delegated member of the research team at a study site
* Any other reason that the Investigator considered made the participant unsuitable to participate
* Participants with no knowledge of their family history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of a GMP SARS-CoV-2 EG.5.1 variant challenge virus in vaccinated healthy adult volunteers with or without previous infection and establish the attack rate (target 50-70%) with optimised dose and screening criteria. | 28 Days
  To assess the safety of a GMP SARS-CoV-2 EG.5.1 variant challenge virus in vaccinated healthy adult volunteers with or without previous infection and establish the attack rate (target 50-70%) with optimised dose and screening criteria.
  To assess safety and human clinical response to SARS-CoV-2 Omicron EG.5.1 intranasal challenge in both previously infected (unvaccinated or vaccinated) and uninfected vaccinated volunteers.
  To evaluate the safety of Omicron variant SARS-CoV-2 challenge in healthy participants, by assessing:
  • Occurrence of AEs within 28 days post-viral challenge (Day 0 to Day 28)
To assess the safety of a GMP SARS-CoV-2 EG.5.1 variant challenge virus in vaccinated healthy adult volunteers with or without previous infection and establish the attack rate (target 50-70%) with optimised dose and screening criteria. | 180 Days
  To assess the safety of a GMP SARS-CoV-2 EG.5.1 variant challenge virus in vaccinated healthy adult volunteers with or without previous infection and establish the attack rate (target 50-70%) with optimised dose and screening criteria.
  To assess safety and human clinical response to SARS-CoV-2 Omicron EG.5.1 intranasal challenge in both previously infected (unvaccinated or vaccinated) and uninfected vaccinated volunteers
  To evaluate the safety of Omicron variant SARS-CoV-2 challenge in healthy participants, by assessing:
  • • Occurrence of SAEs related to the viral challenge (Day 0 to Day 180)
Selection of the SARS-CoV-2 Omicron EG.5.1 dose(s) required to induce upper respiratory tract infection in 50-75% of previously SARS-CoV-2 infected and uninfected vaccinated volunteers (vaccinated or unvaccinated) healthy volunteers following intranasal | 10 Days
  Selection of the SARS-CoV-2 Omicron EG.5.1 dose(s) required to induce upper respiratory tract infection in 50-75% of previously SARS-CoV-2 infected and uninfected vaccinated volunteers (vaccinated or unvaccinated) healthy volunteers following intranasal challenge.
  Laboratory confirmed infection is defined as: two quantifiable (≥LLOQ) RT-PCR measurements from mid turbinate or throat samples, reported on 2 or more consecutive timepoints, starting from Day 2 (inclusive) post-inoculation and up to discharge from quarantine (Day 8 for uninfected participants or Day 10 for infected participants)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, BMBCh FRCP FRCPath PhD, Principal Investigator — Imperial College London